CLINICAL TRIAL: NCT01855854
Title: A Phase II, Prospective Study for Icotinib in Esophageal Carcinoma Patients With EGFR Overexpression or Positive FISH as Second-line Treatment
Brief Title: Second-line Treatment With Icotinib in Esophageal Carcinoma Patients With EGFR Overexpression (IHC 3+) or Positive FISH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-036
Record Dates: First submitted 2013-05-13; First posted 2013-05-17 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib (Experimental): Icotinib: 250 mg is administered orally three times per day, until disease progression or unacceptable toxicity.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Icotinib: 250 mg is administered orally three times per day, until disease progression or untolerable toxicity.
  Other Names: Conmana; BPI-2009

SUMMARY:
This study is designed to evaluate the efficacy and safety of icotinib in treating advanced carcinoma of the gastroesophageal junction and esophagus with EGFR overexpression (IHC 3+) or positive FISH, the primary endpoint is objective response rates.

DETAILED DESCRIPTION:
Epidermal growth factor receptor (EGFR) signaling is critical for cancer cell proliferation, invasion, metastasis, and resistance to apoptosis.EGFR is overexpressed in many epithelial malignancies and therefore makes an attractive therapeutic target.This study is designed to evaluate the efficacy and safety of icotinib in treating advanced carcinoma of the gastroesophageal junction and esophagus with EGFR overexpression (IHC 3+) or positive FISH, the primary endpoint is objective response rates. Secondary endpoints include progress-free survival, overall survival, safety and so on.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic or cytologic diagnosis of carcinoma of the gastroesophageal junction or esophagus;
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria;
* Overexpression of EGFR defined by immunohistochemistry (3+) or gene amplification by fluorescence in-situ hybridisation;
* Have progressed after one chemotherapy regimen;
* Age 18-75 years old with performance status of 0 to 2

Exclusion Criteria:

* Prior targeted therapy with erlotinib, gefitinib, and so on
* Evidence of clinically active Interstitial Lung Diseases (Patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded).
* Known severe hypersensitivity to icotinib or any of the excipients of this product.
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2016-01-07 (Actual)

PRIMARY OUTCOMES:
Objective response rates | 2 months
  Number of participants who achieve complete response or partial response. Either complete response (CR) or partial response (PR) will be evaluated by RECIST, confirmed at least 28 days following the date of the initial response.

SECONDARY OUTCOMES:
Progression Free Survival | 5 months
  A duration from randomization date to disease progression(as defined by RECIST) or death. If a participant are known to have progressed, the time to progression is defined as the time from the date of randomization to the date of progression. Otherwise, a participant will be censored at the last date they are known not to be progressed.
Overall survival | 9 months
  Overall Survival is assessed via calculation of the time to death due to any cause. If a participant is known to have died, the time to death is defined as the time from the date of randomization to the date of death. Otherwise, a participant will be censored at the last date they are known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Sun, MD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jing Huang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Huang J, Fan Q, Lu P, Ying J, Ma C, Liu W, Liu Y, Tan F, Sun Y. Icotinib in Patients with Pretreated Advanced Esophageal Squamous Cell Carcinoma with EGFR Overexpression or EGFR Gene Amplification: A Single-Arm, Multicenter Phase 2 Study. J Thorac Oncol. 2016 Jun;11(6):910-7. doi: 10.1016/j.jtho.2016.02.020. Epub 2016 Mar 12. PMID 26980473